CLINICAL TRIAL: NCT00986921
Title: Mifepristone vs. Laminaria Insertion for Cervical Preparation Prior to Surgical Abortion at 14-16 Weeks
Brief Title: Mifepristone Versus Laminaria Insertion for Cervical Preparation Prior to Surgical Abortion at 14-16 Weeks
Acronym: SAMi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Lynn Borgatta, Principal investigator, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAMi
Record Dates: First submitted 2009-09-23; First posted 2009-09-30 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2013-12

CONDITIONS: Abortion
Keywords: Length of time for procedure to be completed; Need for additional dilation; Subject satisfaction with procedure
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mifepristone (Experimental): women in the mifepristone are would take mifepristone 200 mg for cervical preparation the day before their procedure, and not have dilators inserted. In this group, the sstandard procedure of osmotic dilator insertion is NOT performed.
  Interventions: Drug: mifepristone 200 mg
- Osmotic dilator insertion (Active Comparator): Women assigned to this arm would have the standard procedure for cervical preparation, which is insertion of osmotic dilators the day before the abortion procedure
  Interventions: Device: osmotic dilator insertion

INTERVENTIONS:
Drug: mifepristone 200 mg — mifepristone would be given the day before the procedure
  Arms: mifepristone
Device: osmotic dilator insertion — osmotic dilators (3-6) would be inserted as usual the day before the procedure
  Arms: Osmotic dilator insertion

SUMMARY:
Women who are requesting pregnancy termination at 14-16 weeks, who would normally have osmotic dilator insertion the day before their procedure, would be asked if they wanted to participate. Participants would be randomized to two groups: first, dilator insertion as usual, or second, mifepristone taken the day before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-45 having pregnancy termination at 14-16 weeks

Exclusion Criteria:

* multiple gestation, pre-existing infection, contraindication to osmotic dilators, unable to obtain proper consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L B, MD, MPH, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Borgatta L, Roncari D, Sonalkar S, Mark A, Hou MY, Finneseth M, Vragovic O. Mifepristone vs. osmotic dilator insertion for cervical preparation prior to surgical abortion at 14-16 weeks: a randomized trial. Contraception. 2012 Nov;86(5):567-71. doi: 10.1016/j.contraception.2012.05.002. Epub 2012 Jun 6. PMID 22682721

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the abortion clinic, after they had already consented to the abortion procedure, October 2009 to March 2011.
Pre-assignment Details: All women enrolled were assigned to groups. Group assignment was done very shortly after enrollment.
Groups:
- Standard Osmotic Dilator Insertion: Women assigned to this arm would have the standard procedure, which is insertion of osmotic dilators the day before the procedure.
  Osmotic dilator insertion : osmotic dilators (3-6) would be inserted as usual the day before the procedure.
  All women would have the surgical abortion procedure done on the day following osmotic dilator insertion by standard surgical technique.
- Mifepristone: Women in the mifepristone are would take mifepristone 200 mg the day before their procedure, and not have dilators inserted
  Mifepristone 200 mg : mifepristone would be given the day before the procedure
  All women would have the surgical abortion procedure done on the day following mifepristone, by standard surgical technique.
Period: Overall Study
Arm/Group | Standard Osmotic Dilator Insertion | Mifepristone
Started | 25 | 25
Completed | 24 | 25
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Osmotic Dilators: Women assigned to this arm would have the standard procedure, which is insertion of osmotic dilators the day before the procedure.
  Osmotic dilator insertion : osmotic dilators (3-6) would be inserted as usual the day before the procedure.
  All women would have the surgical abortion procedure done on the day following osmotic dilator insertion by standard technique.
- Mifepristone: Women in the mifepristone are would take mifepristone 200 mg the day before their procedure, and not have dilators inserted
  Mifepristone 200 mg : mifepristone would be given the day before the procedure
  All women would have the surgical abortion procedure done on the day following osmotic dilator insertion by standard technique.
- Total: Total of all reporting groups
Arm/Group | Standard Osmotic Dilators | Mifepristone | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (6) | 24 (5) | 25 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Time for Completion of Procedure
Description: Minutes, from the time of the start of the procedure (speculum insertion) to the conclusion of the procedure (speculum removal)
Time Frame: Performance and completion of the abortion procedure takes 10-20 minutes. The length of the procedure is measured. The procedure occurs approximately 24 hours after enrollment.
Population: Of the 25 women enrolled in the osmotic dilator group, all had osmotic dilators insertion. One woman aborted spontaneously before the surgical abortion; therefore she did not have an abortion procedure and time could not be obtained. she did contribute information about her experience to that point.
Measure: Mean (95% Confidence Interval); unit: Minutes
Groups:
- Mifepristone: Women in the mifepristone are would take mifepristone 200 mg the day before their procedure, and not have dilators inserted. No osmotic dilators are used.
  Mifepristone 200 mg : mifepristone would be given the day before the procedure
  All women would have the surgical abortion procedure done on the day following osmotic dilator insertion by standard technique.
Arm/Group | Standard Osmotic Dilators | Mifepristone
Number analyzed (Participants) | 24 | 25
Minutes | 8.0 [6.75 to 11.47] | 9.87 [8.93 to 11.36]
Statistical Analysis 1: Comparison: Standard Osmotic Dilators vs Mifepristone; Test type: Superiority or Other; p = 0.05, t-test, 1 sided; Data was not distributed normally. After log transformation, the log values were distributed normally; Mean Difference (Final Values) = 1.87, 95% CI 2-sided [0 to 3]

2. Secondary Outcome: Assessment of Ease of Procedure by Operator
Description: The operator for each procedure rated the ease of procedure on a categorical scale. The categories were collapsed into two: "easy or very easy" and "average or difficult".
Time Frame: It is administered shortly after the primary outcome, which is one day after enrollment. The study is complete at that point.
Population: All participants with a completed abortion procedure were rated by the operator as to ease of completing the procedure. The number of women in each group having an abortion procedure rated "easy or very easy" is tabulated
Measure: Number; unit: percentage of participants
Groups:
- Standard Osmotic Dilators: Women assigned to this arm would have the standard procedure, which is insertion of osmotic dilators the day before the procedure.
- Mifepristone: Women in the mifepristone are would take mifepristone 200 mg the day before their procedure, and not have dilators inserted
Arm/Group | Standard Osmotic Dilators | Mifepristone
Number analyzed (Participants) | 24 | 25
percentage of participants | 46 | 36
Statistical Analysis 1: Comparison: Standard Osmotic Dilators vs Mifepristone; The null hypothesis was that the groups would vary, with a p values of less than 0.05; Test type: Superiority or Other; p = 0.49, Chi-squared — A threshold value of p of 0.05 was considered significant

3. Secondary Outcome: Moderate or Severe Pain Overnight
Description: Women wer asked to rank their amount of pain on a catergorical scale. The outcome measure is the number of women experiencing moderate or severe pain overnight (after mifepristone or osmotic dilators, and before the abortions procedure)
Time Frame: Overnight
Population: All participants are included
Measure: Number; unit: percentage of participants
Arm/Group | Standard Osmotic Dilators | Mifepristone
Number analyzed (Participants) | 25 | 25
percentage of participants | 52 | 8
Statistical Analysis 1: Comparison: Standard Osmotic Dilators vs Mifepristone; Test type: Superiority or Other; p = 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Standard Osmotic Dilators | Mifepristone
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
This study was completed as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No